CLINICAL TRIAL: NCT00120575
Title: Hemofiltration for Respiratory Failure Following Hematopoietic Stem Cell Transplantation
Brief Title: Hemofiltration for Respiratory Failure After Bone Marrow Transplantation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT CVVH
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Bone Marrow Transplantation; Respiratory Insufficiency
Keywords: Hemofiltration; Pediatrics
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Hemofiltration

INTERVENTIONS:
Procedure: hemofiltration

SUMMARY:
For children undergoing bone marrow transplantation, respiratory failure is a devastating complication, with mortality expectations well above 60%. The researchers have devised a novel strategy that may greatly improve survival. Hemofiltration, a continuous form of dialysis, was designed as a therapy for critically ill patients with kidney failure. A semi-permeable membrane removes plasma water and solutes (up to about 35,000 Daltons molecular weight). The researchers have treated immuno-compromised children with respiratory failure with hemofiltration. Many inflammatory molecules are of a size well below the limit of the filter. Hemofiltration might remove a critical amount of this inflammatory material, attenuating the unregulated inflammatory response that is central to the development of respiratory failure and progression to multiple organ failure and death. The researchers are conducting a multi-center trial of early continuous hemofiltration for respiratory failure in children following bone marrow transplantation. The researchers will analyze blood and ultrafiltrate using sensitive proteomic methods to detect several inflammatory biochemicals known to be active in this disease, looking for evidence that early active hemofiltration alters the inflammatory response. The researchers will test whether 'early' hemofiltration produces greater survival from respiratory failure in this vulnerable population.

DETAILED DESCRIPTION:
For children undergoing bone marrow transplantation, respiratory failure carries mortality expectations well above 60%. The researchers have published preliminary evidence that continuous hemofiltration may greatly improve survival, if filtration is begun when the child first fulfills clinical criteria for ARDS. This is a departure from standard practice, as hemofiltration is usually begun later in the course (if at all) when multiple organ failure is entrenched. Hemofiltration, a 'renal replacement therapy' for critically ill patients, is a slow, continuous process in which a semi-permeable membrane removes plasma water and solutes (up to about 35 kiloDaltons). Many cytokine and chemokine molecules are smaller than the molecular weight limit of the filter; hemofiltration might remove a critical amount, attenuating the unregulated inflammatory response responsible for respiratory failure and progression to multiple organ failure and death. The researchers will conduct a multi-center randomized trial assessing the effect of hemofiltration on survival from respiratory after bone marrow (or more precisely, hematopoietic stem cell) transplantation. The researchers will perform sensitive proteomic assays of serum and ultrafiltrate, to detect the presence of cytokines and chemokines known to be active in idiopathic pneumonia syndrome. Resulting profiles will constitute a uniquely complex description of ultrafiltrate and may provide evidence for modulation of immune function by hemofiltration.

ELIGIBILITY:
Inclusion Criteria:

* hematopoietic stem cell recipient
* respiratory failure fulfilling ARDS criteria
* mechanical ventilation (invasive / non-invasive)

Exclusion Criteria:

* extracorporeal membrane oxygenation (ECMO)
* predominance of congestive heart failure
* code status: a patient must be willing to accept invasive mechanical ventilation if clinically indicated

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112
Dates: Start 2005-01; Study Completion 2008-09

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
PELOD organ failure score
number of ventilator-free days
duration of hospitalization
functional outcome score

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V DiCarlo, MD, Principal Investigator — Stanford University
Locations (7):
- United States (4):
  - Children's Hospital and Research Center, Oakland, California
  - Children's Healthcare of Atlanta @ Egleston, Atlanta, Georgia
  - Duke University, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Children's Hospital of British Columbia, Vancouver, British Columbia, Canada
- University of Ulm, Ulm, Germany
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Background] DiCarlo JV, Alexander SR, Agarwal R, Schiffman JD. Continuous veno-venous hemofiltration may improve survival from acute respiratory distress syndrome after bone marrow transplantation or chemotherapy. J Pediatr Hematol Oncol. 2003 Oct;25(10):801-5. doi: 10.1097/00043426-200310000-00012. PMID 14528104
- [Background] Di Carlo JV, Alexander SR. Hemofiltration for cytokine-driven illnesses: the mediator delivery hypothesis. Int J Artif Organs. 2005 Aug;28(8):777-86. doi: 10.1177/039139880502800803. PMID 16211527